CLINICAL TRIAL: NCT04223830
Title: Initial Case Series With Exalt Single-Use Duodenoscope - Expanded User Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E7158
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Exalt DScope 01B (Experimental): Subjects will have a clinically indicated per standard of care endoscopic retrograde cholangiopancreatography (ERCP) or other duodenoscope-based procedure performed using the Exalt single use duodenoscope study device. Subjects are considered enrolled after completing the study specific informed consent form.
  Interventions: Device: Exalt Model D Single-Use Duodenoscope

INTERVENTIONS:
Device: Exalt Model D Single-Use Duodenoscope — Subjects will have a clinically indicated per standard of care endoscopic retrograde cholangiopancreatography (ERCP) or other duodenoscope-based procedure performed with the Exalt single use duodenoscope study device.

SUMMARY:
The objective of this study is to confirm procedural performance of the Exalt Model D Single-Use Duodenoscope in Endoscopic Retrograde Cholangio-Pancreatography (ERCP) and other duodenoscope-based procedures.

DETAILED DESCRIPTION:
The main objective of this study to confirm the design and operating specifications of the Exalt Model D Single-Use Duodenoscope in Endoscopic Retrograde Cholangio-Pancreatography (ERCP) and other duodenoscope-based procedures in study subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Scheduled for a clinically indicated endoscopic retrograde cholangiopancreatography (ERCP)

Exclusion Criteria:

* Altered pancreaticobiliary anatomy
* Potentially vulnerable subjects, including, but not limited to pregnant women
* Subjects for whom endoscopic techniques are contraindicated
* Patients who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
* Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Slivka, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (7):
- United States (6):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data, analytic methods, and study materials for this study may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

REFERENCES:
- [Derived] Slivka A, Ross AS, Sejpal DV, Petersen BT, Bruno MJ, Pleskow DK, Muthusamy VR, Chennat JS, Krishnamoorthi R, Lee C, Martin JA, Poley JW, Cohen JM, Thaker AM, Peetermans JA, Rousseau MJ, Tirrell GP, Kozarek RA; EXALT Single-use Duodenoscope Study Group. Single-use duodenoscope for ERCP performed by endoscopists with a range of experience in procedures of variable complexity. Gastrointest Endosc. 2021 Dec;94(6):1046-1055. doi: 10.1016/j.gie.2021.06.017. Epub 2021 Jun 26. PMID 34186052

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 208 patients provided informed consent for the study, however prior to participation 8 patients were subsequently found to be ineligible and are considered screen failures per protocol.
Groups:
- Exalt DScope 01B: Subjects will have a clinically indicated per standard of care ERCP or other duodenoscope-based procedure performed using the Exalt single use duodenoscope study device. Subjects are considered enrolled after completing the study specific informed consent form.
  Exalt Model D Single-Use Duodenoscope: Subjects will have a clinically indicated per standard of care ERCP or other duodenoscope-based procedure performed with the Exalt single use duodenoscope study device.
Period: Overall Study
Arm/Group | Exalt DScope 01B
Started | 200
Completed | 190
Not Completed | 10
Not completed — Lost to Follow-up | 9
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exalt DScope 01B
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 10
  United States | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Endoscopic Retrograde Cholangiopancreatography (ERCP) Procedure
Description: The ability to complete the ERCP procedure for the intended indication(s); outcome reported as "success" or "failure".
  Examples include but are not limited to: biliary stent placement, pancreatic stent placement, sphincterotomy, and clearance of bile duct stones.
Time Frame: Procedure success is assessed at the end of the procedure (within 24 hours on study day 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Exalt DScope 01B
Number analyzed (Participants) | 200
Participants | 193

2. Secondary Outcome: Endoscopist Overall Satisfaction Rating of the Exalt Single-use Duodenoscope
Description: Endoscopist overall satisfaction rating of the Exalt single-use duodenoscope, as compared to their past experience with marketed reusable duodenoscopes. The overall satisfaction rating is recorded on a scale of 1 (unsatisfied) to 10 (very satisfied), with 1 being the minimum value (worse) and 10 being the maximum value (better). A rating of 1 indicates the endoscopist is unsatisfied with the Exalt single-use duodenoscope, as compared to past experience with marketed reusable duodenoscopes. A rating of 10 indicates the endoscopist is very satisfied with the Exalt single-use duodenoscope, as compared to past experience with marketed reusable duodenoscopes.
Time Frame: Endoscopists will rate their experience with the Exalt single-use duodenoscope immediately following the completion of the study procedure on study day 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Exalt DScope 01B: Overall satisfaction
Arm/Group | Exalt DScope 01B
Number analyzed (Participants) | 200
score on a scale | 7.6 (2.1)

3. Secondary Outcome: Number of Participants With Crossover From Exalt Single-use Duodenoscope to Reusable Duodenoscope
Description: The need to use a reusable duodenoscope for any task which cannot be adequately performed with the Exalt single-use duodenoscope is considered a crossover.
Time Frame: Crossover is monitored throughout the procedure (within 24 hours on study day 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Exalt DScope 01B
Number analyzed (Participants) | 200
Participants | 19

4. Secondary Outcome: Number of Serious Adverse Events (SAEs) Related to the Device and/or the Procedure
Description: Number of serious adverse events (SAEs) related to the device and/or the procedure.
Time Frame: SAEs are assessed through 7 days after the procedure.
Measure: Number; unit: Related Serious Adverse Events
Arm/Group | Exalt DScope 01B
Number analyzed (Participants) | 200
Related Serious Adverse Events | 15

ADVERSE EVENTS:
Time Frame: Occurrence of adverse events were collected through 7 days (+/- 2 days) after the index procedure.
Description: All adverse events were collected, regardless of relationship to study device and/or procedure. Given the nature of the study procedure, any crossover between the Exalt single-use duodenoscope and the reusable duodenoscope would have occurred during the same study procedure therefore, it is difficult to determine the relatedness of adverse events to the Exalt single-use duodenoscope or to the reusable duodenoscope. Adverse events are therefore reported in a combined fashion.
Arm/Group | Exalt DScope 01B
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 13/200
Other Adverse Events (participants affected / at risk) | 20/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exalt DScope 01B (N=200)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Oesophageal mucosal tear (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exalt DScope 01B (N=200)
Abdominal Pain (Gastrointestinal disorders) | 8 (8)
Pancreatitis (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT04223830/Prot_SAP_002.pdf